CLINICAL TRIAL: NCT07261982
Title: Efficacy of Pressure Pad vs Pressure Bandage Immobilisation for Snake Bite First Aid in Healthy Volunteers.
Brief Title: Analysis of the Efficacy of Pressure Pad vs Pressure Bandage Immobilisation for Snake Bite First Aid in Healthy Volunteers.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Townsville University Hospital (Other)
Responsible Party: Principal Investigator, Adam Holyoak, Senior Staff Specialist, Townsville University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EMLE-280R41-2024-HOLYOAK
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Snake Bites; Snakebite; Snake Envenomation; Snake Bite; First Aid
Keywords: Snakebite; First aid; Pressure bandage immobilisation; Pressure pad
MeSH Terms: conditions — Snake Bites

STUDY DESIGN:
Intervention Model Description: Data analysis will be undertaken by the research team which includes a biostatistician. For a standard two-period, two-sequence cross-over design, the investigators anticipate a sample size of N=24 will achieve 91% power at a 5% significance level assuming the absolute difference between the two-treatment means is 1 minute and the within-subject standard deviation is 1 minute. This will allow detection of significant differences between all interventional scans and controls and determine the efficacy of each first aid technique. A >90% power has been chosen due to the paucity of data in the literature to guide better predict effect size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of control, pressure bandage immobilisation and pressure pad first aid techniques (Experimental): Each subject will be injected with mock venom in either their hand or foot and then either no first aid (control), pressure bandage immobilisation, or pressure pad first aid techniques will be applied. The passage of mock venom (Technetium-99m sulphur colloid) through the subject's lymphatic system will be tracked by nuclear medicine imaging. Each subject will undergo repeated scans each using a different location/first aid method so that all subjects will have data on all six possible permutations in a randomised order. Time in seconds for the mock venom to travel to regional lymph nodes in the relevant limb will be recorded and compared across the different first aid techniques.
  Interventions: Other: Pressure bandage immobilisation first aid; Other: Pressure pad first aid; Other: Control - no first aid

INTERVENTIONS:
Other: Pressure bandage immobilisation first aid — Pressure Bandage Immobilisation Technique (PBI):
  1. An elastic bandage of 100mm width will be applied to the full length of the involved limb, starting from the fingers or toes and moving proximally until the whole limb is bandaged, bandaging over clothing if required.
  2. The desired pressure of the bandage (~60mmHg) will be obtained by utilising "smart" bandages which have special markings that take on the shape of a square when the bandage is applied at this pressure/tension. Prior to use on each subject, the accuracy of this process will be confirmed via pressure manometry using an infant blood pressure cuff bladder placed under the wraps of the elastic bandage and connected to a manometer as per Canale et al.
  3. Splinting of the limb will be performed using a sling for the arm, and a wooden splint for the leg.
Other: Pressure pad first aid — Pressure Pad Technique (PP):
  1. A square gauze pad of 5 sheets thickness with an overall size of 80x80mm will be applied to the injection site.
  2. The gauze pad will be secured using an elastic bandage of 100mm width at a tension of ~60mmHg using a "smart" bandage. Prior to use on each subject, the accuracy of this process will be confirmed via pressure manometry using an infant blood pressure cuff bladder placed under the wraps of the elastic bandage and connected to a manometer as per Canale et al.
  3. Splinting of the limb will be performed using a sling for the arm, and a wooden splint for the leg.
Other: Control - no first aid — Control (no first aid technique applied):
  1. Imaging will be done with the subject lying supine and still without the application of either bandaging technique
  2. Splinting of the limb will be performed using a sling for the arm, and a wooden splint for the leg.

SUMMARY:
Snake bite affects thousands of Australians every year, but few die as a result due to high quality first aid and timely medical care. Good first aid should be simple, standardised, use minimal or readily available equipment, and be able to be utilised effectively with no or minimal training by the rescuer. Over time the first aid methods used to manage snake bite in Australia have been questioned due to issues with efficacy, and some emerging evidence of harm from their use. There is little experimental data in the literature to support current first aid practices, and what exists suggests further research is required. This study aims to examine and compare the effectiveness of two first aid methods by tracking the movement of a mock venom through the body when each first aid method is used. This will provide important information about the suitability of current techniques used in Australia and whether a proposed simpler alternative technique is as effective. Currently, initial treatment of snake bite involves early first aid with the application of a pressure bandage and immobilisation (PBI) of the limb. There is limited data to support the basis of this technique and emerging evidence of harm when applied incorrectly. This project sets out to evaluate PBI compared to another technique involving the application of a pressure pad (PP) at the bite site (which is easier to do, and used in many countries outside of Australia). The project aims to determine whether each technique is effective, and whether the PP technique is at least as effective as PBI. To do this 24 participants will be recruited to undergo study with mock venom injected into their hand or foot and having either PBI or PP applied. The mock venom will then be traced with a gamma camera to determine rate of flow through the lymphatic system, which is how venom travels in the body. It is expected that the project will demonstrate the efficacy of both techniques, and that the PP will be at least as effective as PBI. This will provide a basis for change in the current first aid recommendations for snake bite first aid in Australia, and improve the care provided.

DETAILED DESCRIPTION:
Snake bite affects over 5 million people worldwide each year, with between 80000 and 137000 deaths. In Australia there are over 10000 snake bites annually, with over one third of these resulting in envenomation. Of those envenomed, only 2 to 4 die each year since the development of antivenom and the institution of appropriate first aid.

The current standard of first aid for snake bite in Australia is the application of the Pressure Bandage Immobilisation (PBI) technique that was originally described by Sutherland et al. in 1979. However, since the development of this technique there has been critique and debate in the medical literature surrounding the actual efficacy of the method when applied in the field. Much of this critique centred around inappropriate application of the technique, insufficient pressure in the application of the bandage, or lack of immobilisation. Despite the popularity of PBI technique, there are still large numbers of patients presenting with snake bite without having any first aid applied at all. Retrospective analysis by some of the original publication by Sutherland has also called into question the validity of the technique itself. Yet, with the inception of PBI and antivenom, the number of snake bite deaths in this country has decreased significantly. As such the technique has been promulgated without much question and remains the recommended method of snake bite first aid in Australia by the Australian Resuscitation Council (ARC). Recently however, there have been calls for more robust research into snake bite first aid, especially with growing evidence of harm (including ineffective compression, pressure injury, nerve injury, limb amputation etc) that is likely the direct result of incorrect application of the PBI technique. The key principles of first aid are to preserve life, prevent deterioration and promote recovery. One of the key objectives of the ARC is to promote simplicity and uniformity in techniques used in resuscitation.

Australian venomous snakes of medical significance all come from the family Elapidae, which are not known for a strong localised tissue effect from their venom. This in is contrast to other countries who also have venomous snakes from the Viperidae family whose venoms often contain strongly myotoxic and locally necrotic venom components. As such, the PBI technique has largely been avoided in locations outside Australia due to concerns for compartmentalisation of necrotoxic and myotoxic venom worsening localised effects. Promising data has emerged from research in Myanmar that supports the use of a more localised Pressure Pad (PP) or "Monash method" technique (which is popular in many areas outside Australia) that is simpler to apply correctly, less likely to cause injury to the patient, and as such may be superior to the current PBI method for Australian snake bite first aid. Most notably for the PP technique, data from its use in envenomated patients does not indicate an increase in local tissue effects, even in venoms containing high proportions of myotoxic and necrotoxic components. A further advantage of the PP technique is that can be applied to bites on the torso or abdomen, which is not the case for the PBI technique.

The underlying mechanism of PBI as proposed by Sutherland is that the bandage be applied at such a pressure to arrest flow within the lymphatic system (in most Australian snake bites, venom is injected subcutaneously and transported through the body in the lymphatic system) allowing more time for the victim to receive medical attention and antivenom when indicated. There is reasonable consensus in published research that the required pressure to retard lymphatic flow is between approximately 50-70mmHg. Such pressure can be delivered in the PBI technique using elasticised bandages wrapped over the entire length of the affected limb, the limb then being immobilised with a splint. The PP technique as published may create a higher pressure at the site of the pad, but is only applied locally, rather than to the whole limb, again with splinting to facilitate immobilisation. Importantly, for both methods, immobilisation of the limb along with the specific bandaging technique is necessary to affect a slowing of the travel of venom. This project seeks to examine the efficacy of both the PBI and PP techniques and determine whether the PP technique is at least equivalent to the PBI method as first aid, especially when using a regulated pressure of approximately 60mmHg.

Should the data from this project demonstrate the efficacy of the PP technique, given its relative simplicity, less likelihood of causing deleterious effects to the patient, and uniformity with first aid techniques used elsewhere in the world, it would give reason for the ARC to re-consider its recommended first aid treatment in Australia. An easy to use technique would also likely result in more victims of snake bite having appropriate first aid applied which may again reduce the progression of envenomation symptoms that if untreated require longer hospital lengths of stay. Also, preventing harm from incorrectly applied first aid techniques is important in reducing morbidity associated with snake bite.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or greater
* No known or clinically evident lymphatic condition (eg. lymphoedema, lymph node surgery etc)
* No known cardiac failure
* No known peripheral vascular disease
* No known renal or hepatic impairment
* No known lymphoma

Exclusion Criteria:

* Age less than 18 years old
* Pregnant
* Breast feeding
* Allergy to Technetium-99m sulphur colloid
* Presence of any of the conditions mentioned in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Time for mock venom to reach regional lymph nodes following injection | From the date of enrolment until all scans are completed (minimum of 12 weeks, maximum of 18 months).
  Time (in seconds) will be recorded from the injection of Tn-99m sulfur colloid until signal is detected at the regional lymph nodes for the relevant limb, and then until there is evidence of entry to the systemic circulation (as demonstrated by signal detection in the liver). Times will be judged by the reporting radiologist on the basis of the time stamp on the relevant image relating to signal detection at the relevant location. Each scan will run for up to 30 minutes, with intervention scans having the first aid technique removed at this point and running for a further 30 minutes. This allows demonstration of movement of mock venom through the lymphatic system after removal of first aid if the initial application of first aid is efficacious enough to completely retard mock venom movement. Distance from injection site to either groin or axilla (as relevant) will also be measured at each scan so that a lymphatic flow rate is able to be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Adam L Holyoak, Principal Investigator — Townsville University Hospital; Mark Little, Principal Investigator — Cairns Hospital; Tyson Reeve, Principal Investigator — Queensland X-Ray; Jade Bax, Principal Investigator — Queensland X-Ray; Theophilus I Emeto, Principal Investigator — James Cook University, Queensland, Australia
Locations (1):
- Queensland X-Ray, Hyde Park, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be provided on request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be provided on request upon completion of the study and will be available for up to 10 years following completion of the study.
  Supporting information will be available as or when available until 10 years following completion of the study.
Access Criteria: Parties wishing to access the IPD will be able to do so by contacting the primary author of the study, and will be provided with the relevant data etc as required

REFERENCES:
- [Background] Sutherland SK. The pressure immobilisation technique. Med J Aust. 1994 Dec 5-19;161(11-12):700-1. No abstract available. PMID 7830642
- [Background] Smith H. Uptake of "mock-venom". Med J Aust. 1982 Jul 24;2(2):66
- [Background] Anker RL, Straffon WG, Loiselle DS, Anker KM. Snakebite. Comparison of three methods designed to delay uptake of 'mock venom'. Aust Fam Physician. 1983 May;12(5):365-8. PMID 6351824
- [Background] Pe T, Mya S, Myint AA, Aung NN, Kyu KA, Oo T. Field trial of efficacy of local compression immobilization first-aid technique in Russell's viper (Daboia russelii siamensis) bite patients. Southeast Asian J Trop Med Public Health. 2000 Jun;31(2):346-8. PMID 11127337
- [Background] Tun-Pe, Aye-Aye-Myint, Khin-Ei-Han, Thi-Ha, Tin-Nu-Swe. Local compression pads as a first-aid measure for victims of bites by Russell's viper (Daboia russelii siamensis) in Myanmar. Trans R Soc Trop Med Hyg. 1995 May-Jun;89(3):293-5. doi: 10.1016/0035-9203(95)90547-2. PMID 7660439
- [Background] Little M. Harm due to the use of pressure bandage immobilisation in patients bitten by snakes in Australia. Clin Toxicol (Phila). 2023 Aug;61(8):611-612. doi: 10.1080/15563650.2023.2252586. Epub 2023 Sep 5. PMID 37668172
- [Background] Pressure/immobilisation first aid treatment of snake bite. Med J Aust. 1982 Feb 20;1(4):155, 157. No abstract available. PMID 7078485
- [Background] Pearn JH, Morrison JJ, Charles NT. First aid in snake bite; comment on mock venom. Med J Aust. 1982 Jul 24;2(2):65-6. doi: 10.5694/j.1326-5377.1982.tb124243.x. No abstract available. PMID 7121362
- [Background] Parker-Cote J, Meggs WJ. First Aid and Pre-Hospital Management of Venomous Snakebites. Trop Med Infect Dis. 2018 Apr 24;3(2):45. doi: 10.3390/tropicalmed3020045. PMID 30274441
- [Background] Anker RL, Straffon WG, Loiselle DS, Anker KM. Retarding the uptake of "mock venom" in humans: comparison of three first-aid treatments. Med J Aust. 1982 Mar 6;1(5):212-4. doi: 10.5694/j.1326-5377.1982.tb132272.x. PMID 7087836
- [Background] Sutherland SK, Coulter AR, Harris RD. Rationalisation of first-aid measures for elapid snakebite. Lancet. 1979 Jan 27;1(8109):183-5. doi: 10.1016/s0140-6736(79)90580-4. PMID 84206
- [Background] Rogers IR, Winkel KD. Struan Sutherland's "Rationalisation of first-aid measures for elapid snakebite"--a commentary. Wilderness Environ Med. 2005 Fall;16(3):160-3. doi: 10.1580/er20-04.1. No abstract available. PMID 16209471
- [Background] Currie BJ, Canale E, Isbister GK. Effectiveness of pressure-immobilization first aid for snakebite requires further study. Emerg Med Australas. 2008 Jun;20(3):267-70. doi: 10.1111/j.1742-6723.2008.01093.x. PMID 18549384
- [Background] Canale E, Isbister GK, Currie BJ. Investigating pressure bandaging for snakebite in a simulated setting: bandage type, training and the effect of transport. Emerg Med Australas. 2009 Jun;21(3):184-90. doi: 10.1111/j.1742-6723.2009.01180.x. PMID 19527277
- [Background] Welton RE, Liew D, Braitberg G. Incidence of fatal snake bite in Australia: A coronial based retrospective study (2000-2016). Toxicon. 2017 Jun 1;131:11-15. doi: 10.1016/j.toxicon.2017.03.008. Epub 2017 Mar 10. PMID 28288937
- [Background] Howarth DM, Southee AE, Whyte IM. Lymphatic flow rates and first-aid in simulated peripheral snake or spider envenomation. Med J Aust. 1994 Dec 5-19;161(11-12):695-700. PMID 7830641
- [Background] Seifert SA, Armitage JO, Sanchez EE. Snake Envenomation. N Engl J Med. 2022 Jan 6;386(1):68-78. doi: 10.1056/NEJMra2105228. PMID 34986287
- [Background] Norris RL, Ngo J, Nolan K, Hooker G. Physicians and lay people are unable to apply pressure immobilization properly in a simulated snakebite scenario. Wilderness Environ Med. 2005 Spring;16(1):16-21. doi: 10.1580/PR12-04.1. PMID 15813142
- [Background] Avau B, Borra V, Vandekerckhove P, De Buck E. The Treatment of Snake Bites in a First Aid Setting: A Systematic Review. PLoS Negl Trop Dis. 2016 Oct 17;10(10):e0005079. doi: 10.1371/journal.pntd.0005079. eCollection 2016 Oct. PMID 27749906
- See also: World Health Organisation. Snakebite envenoming. — https://www.who.int/news-room/fact-sheets/detail/snakebite-envenoming
- See also: Australian Venom Research Unit. FAQ: How common is snakebite in Australia — https://biomedicalsciences.unimelb.edu.au/departments/department-of-biochemistry-and-pharmacology/engage/avru/advice-and-resources/frequently-asked-questions
- See also: Australian Venom Research Unit. The global scale of snakebite. Snakebite envenoming: a neglected tropical disease — https://biomedicalsciences.unimelb.edu.au/departments/department-of-biochemistry-and-pharmacology/engage/avru/discover/snakebite-envenoming-a-neglected-tropical-disease
- See also: 16. Australian Resuscitation Council. Envenomation - pressure immobilisation technique — https://resus.org.au/the-arc-guidelines/
- See also: Australian Resuscitation Council. Aims and objectives of the ARC — https://resus.org.au/aims-and-objectives-of-the-arc/

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT07261982/Prot_SAP_000.pdf
  • Informed Consent Form: Patient Consent Form (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT07261982/ICF_001.pdf
  • Informed Consent Form: Patient Information Form (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT07261982/ICF_002.pdf